CLINICAL TRIAL: NCT06303947
Title: A Randomized Trial to Explore the Effect of Oral Enteral Nutrition Feeding in Parkinson Disease
Brief Title: Effect of Oral Enteral Nutrition Feeding in Parkinson Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IOE-PKS
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oro-esophageal Tube+comprehensive rehabilitation therapy (Experimental): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  The group was given enteral nutritional support with Intermittent Oro-esophageal Tube Feeding
  Interventions: Device: Intermittent Oro-esophageal Tube; Behavioral: Comprehensive rehabilitation training
- Nasogastric Tube+comprehensive rehabilitation therapy (Active Comparator): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Besides, the group was given enteral nutritional support with Nasogastric Tube Feeding according to the relevant guidelines.
  Interventions: Device: Nasogastric tube; Behavioral: Comprehensive rehabilitation training

INTERVENTIONS:
Device: Intermittent Oro-esophageal Tube — The group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure: Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Intermittent Oro-esophageal Tube+comprehensive rehabilitation therapy
Device: Nasogastric tube — The group is given enteral nutritional support with Nasogastric tube according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: Nasogastric Tube+comprehensive rehabilitation therapy
Behavioral: Comprehensive rehabilitation training — Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.

SUMMARY:
The goal of this or clinical trial is to explore Intermittent Oro-esophageal Tube Feeding vs. Nasogastric Tube Feeding on nutritional status, dysphagia, and activities of daily living in patients with Parkinson's disease. The main question it aims to answer are:

• Can stellate ganglion block improve the nutritional status, dysphagia, and activities of daily living in patients with Parkinson's disease, better than Nasogastric Tube Feeding.

Participants will be divided into the control group and observation group evenly. All the patients were provided with routine therapy and given nutritional support by Intermittent Oro-esophageal Tube Feeding and Nasogastric Tube Feeding respectively. The nutritional status, swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

DETAILED DESCRIPTION:
Nasogastric tube feeding has been widely used in patients with Parkinson's disease but has a significant risk of complications. Intermittent Oro-esophageal Tube Feeding is an established enteral nutrition approach that can be used with comprehensive rehabilitation therapy.

The goal of this or clinical trial is to explore Intermittent Oro-esophageal Tube Feeding vs. Nasogastric Tube Feeding on nutritional status, dysphagia, and activities of daily living in patients with Parkinson's disease. The main question it aims to answer are:

• Can stellate ganglion block improve the nutritional status, dysphagia, and activities of daily living in patients with Parkinson's disease, better than Nasogastric Tube Feeding.

Participants will be divided into the control group and observation group evenly. All the patients were provided with routine therapy and given nutritional support by Intermittent Oro-esophageal Tube Feeding and Nasogastric Tube Feeding respectively. The nutritional status, swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Water swallow test> Level 3.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Serum albumin level | day 1 and day 15
  Serum albumin was recorded via blood routine test.(Alb, g/L)
Hemoglobin | day 1 and day 15
  Hemoglobin was recorded via blood routine test.(Hb, mg/L)

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 15
  The activities of daily living was assessed utilizing the Modified Barthel Index (MBI). Modified Barthel Index includes the following 10 subscales. For each subscale, choices encoded with the score 10, 8, 5, 2, 0 are set with the decreasing level of self-dependence, while the final total is positively correlated with Activities of daily living. Cronbach's α of questionnaire adopted is 0.916.
Functional Oral Intake Scale | day 1 and day 15
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No